CLINICAL TRIAL: NCT05227989
Title: Functional and Respiratory Outcomes of Mechanically Ventilated Children in Pediatric Intensive Care, a Prospective Cohort Study
Brief Title: Outcome of Children Post Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Laval University (Other)
Responsible Party: Principal Investigator, Laurence Ducharme-Crevier, Principal Investigator, Pediatric Intensivist, St. Justine's Hospital
Other Study IDs: MP-21-2022-3571
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Post Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation is a life-saving therapy widely used in PICU, but not without adverse effects. The mid-term outcome of mechanically ventilated children who survive critical illness is still poorly defined, in terms of respiratory status, functionality, and quality of life. This lack of knowledge can lead to delays in management and thus hinder the recovery of children.

The aim of this study is to determine the impact on the functional and respiratory outcome of pediatric patients after a stay a PICU of the province of Quebec.

DETAILED DESCRIPTION:
This is a prospective longitudinal cohort study of pediatric patients requiring mechanical ventilation for at least 48 hours, in all 4 PICUs in the province of Quebec (Canada).

In follow-up PICU clinics, children and family outcomes will be evaluated 2, 6 and 12 months post PICU discharge.Children and their families will be enrolled locally from each PICU, their baseline data will be collected by local research staff and their post-discharge outcomes will be followed centrally from the Centre Hospitalier Universitaire Sainte-Justine.

The specific aims are to determine the functional, respiratory and neurocognitive function of PICU survivors and Health related Quality of life. Psychosocial status of the child and parents will also be determined.

The primary goal is to describe the impact of a critical illness and mechanical ventilation on PICU survivors and their families in order to improve the health and well-being of PICU survivors and their families, and ultimately to improve the care of children after a PICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 18 years of age;
* Admission to a PICU at the Centre Hospitalier Universitaire Sainte-Justine (CHUSJ), Montreal Children's Hospital (MCH), Centre Hospitalier Universitaire de Québec - Université Laval (CHUL) or Centre Hospitalier Universitaire de Sherbrooke (CHUS);
* Patients with invasive mechanical ventilation for ≥48 hours.

Exclusion Criteria:

* Patients admitted for congenital heart surgery

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to a PICU requiring mechanical ventilation for at least 48 hours.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Functional status | 12 months
  Functional Status Scale (FSS) Final scores range from 6 to 30 Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Respiratory status | 12 months
  6 minute walk test Result expressed in meters Higher score means better function
Health related Quality of life | 12 months
  PedsQL™ 4.0 Generic Core or Infant Scales (self report or report parent) Final scores range from 0 to 100 Higher scores mean a better outcome
Psychosocial status of the child | 12 months
  Child PTSD Symptom Scale for DSM-5 (CPSS-5) (children 1year+) The total severity score ranges from 0 to 80 Higher scores mean a worse outcome.
Psychosocial status of the parents | 12 months
  Hospital Anxiety & Depression Scale (HADS) (parents) Each category (Anxiety and Depression) range from 0 to 21) Higher scores mean a worse outcome.
Neurocognition | 12 months
  Test according to age of patient:
  Bayley Scales of Infant Development III (1-30months) Wechsler Preschool and Primary Scale of Intelligence IV (WPPSI) (30months-7year) Wechsler Intelligence Scale for Children V (WISC)(7-16year) Wechsler Adult Intelligence Scale IV (WAIS)(16year+) These tests provide standardized norms, percentiles and age equivalent percentiles. The mean score is 100 ± SD15.
  Higher score mean better functioning

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Ducharme-Crevier, MD MSc, Principal Investigator — St. Justine's Hospital
Locations (4):
- Canada (4):
  - CHU Sainte-Justine, Montreal, Quebec
  - Hôpital de Montréal pour enfants (MCH), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Québec - Université Laval (CHUL), Québec